CLINICAL TRIAL: NCT02316197
Title: A Multicenter, Open-Label, Dose-Escalating Phase I Trial of the DNA-PK Inhibitor MSC2490484A in Subjects With Advanced Solid Tumors or Chronic Lymphocytic Leukemia
Brief Title: Clinical Phase I Study Investigating MSC2490484A, an Inhibitor of a DNA-dependent Protein Kinase, in Advanced Solid Tumors or Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR100036-001; 2014-003099-22 (EudraCT Number)
Record Dates: First submitted 2014-12-10; First posted 2014-12-12 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Advanced Solid Tumors; Chronic Lymphocytic Leukemia
Keywords: DNA-PK Inhibitor; Advanced solid tumors; Chronic lymphocytic Leukemia; Phase I, first-in-human; Dose escalation; Dose expansion; Safety profile; Tolerability; PK; Antitumor activity; Maximum tolerated dose; M3814
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — peposertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- MSC2490484A 100 mg QD (Experimental): Participants received MSC2490484A capsules 100 milligram (mg) orally, once daily (QD) from Day 1 to Day 21 of each treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, and/or occurrence of any criterion for withdrawal from study or M3814.
  Interventions: Drug: MSC2490484A (M3814)
- MSC2490484A 200 mg QD (Experimental): Participants received MSC2490484A capsules 200 mg orally, QD from Day 1 to Day 21 of each treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, and/or occurrence of any criterion for withdrawal from study or M3814.
  Interventions: Drug: MSC2490484A (M3814)
- MSC2490484A 150 mg BID (Experimental): Participants received MSC2490484A capsules 150 mg orally, twice daily (BID) from Day 1 to Day 21 of each treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, and/or occurrence of any criterion for withdrawal from study or M3814.
  Interventions: Drug: MSC2490484A (M3814)
- MSC2490484A 200 mg BID (Experimental): Participants received MSC2490484A capsules 200 mg orally, BID from Day 1 to Day 21 of each treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, and/or occurrence of any criterion for withdrawal from study or M3814.
  Interventions: Drug: MSC2490484A (M3814)
- MSC2490484A 300 mg BID (Experimental): Participants received MSC2490484A capsules 300 mg orally, BID from Day 1 to Day 21 of each treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, and/or occurrence of any criterion for withdrawal from study or M3814.
  Interventions: Drug: MSC2490484A (M3814)
- MSC2490484A 400 mg BID (Experimental): Participants received MSC2490484A capsules 400 mg orally, BID from Day 1 to Day 21 of each treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, and/or occurrence of any criterion for withdrawal from study or M3814.
  Interventions: Drug: MSC2490484A (M3814)
- MSC2490484A 400 mg BID RP2D (Experimental): Participants received MSC2490484A capsules 400 mg recommended Phase II dose (RP2D) orally, BID from Day 1 to Day 21 of each treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, and/or occurrence of any criterion for withdrawal from study or M3814.
  Interventions: Drug: MSC2490484A (M3814)

INTERVENTIONS:
Drug: MSC2490484A (M3814) — Participants received MSC2490484A capsules at escalated dose from 100 mg to 400 mg orally from Day 1 to Day 21 of each treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, and/or occurrence of any criterion for withdrawal from study or M3814.
  Other Names: M3814; Peposertib

SUMMARY:
MSC2490484A is an investigational drug that is being evaluated for the treatment of subjects with advanced solid tumors or chronic lymphocytic leukemia (CLL) that likely differs from other cancers in how it repairs damaged DNA (genetic material). This is a first-in-man Phase I study, which means that it is the first time the study drug is being used in humans. The main purpose is to determine the highest dose that does not cause unacceptable side effects. The second is to determine the appropriate dose to use in future research for subjects with cancer. Othergoals of the study are to learn about the drug's safety and side effects, how it affects the tumor, and how the body processes the drug.

DETAILED DESCRIPTION:
This is a Phase I, first-in-human, open-label, dose escalation, and dose expansion trial designed to explore the safety, tolerability, PK and PD profiles, and clinical activity of MSC2490484A administered daily as a single agent to subjects with advanced solid tumors or CLL likely to have alterations in DNA repair mechanisms.

Dose Escalation : Subjects will receive MSC2490484A continuously at the starting dose of 100 mg once daily. Sequential treatment cohorts will receive ascending doses of MSC2490484A once daily or twice daily (if determined to be appropriate by the Safety Monitoring Committee [SMC]) following a standard "3+3" design. The SMC will make dose escalation decisions based on review of available safety, tolerability, Pharmacokinetic (PK), and Pharmacodynamic (PD) data. Once the maximum tolerated dose (MTD) has been established, an Recommended Phase II Dose (RP2D) will be defined by the SMC, either at the MTD level or another dose level, depending on the available data on safety, efficacy, PK, and PD observed in the trial. The SMC may decide to stop dose escalation at any time during the trial.

Up to 12 subjects will be enrolled at the RP2D/Optimal biologic dose (OBD) to confirm safety and tolerability and explore the PK and PD profile of MSC2490484A.

Expansion cohorts: Once subjects have been evaluated at the RP2D, additional subjects will be enrolled into 2 or more expansion cohorts (20 evaluable subjects per expansion cohort) to evaluate clinical efficacy in tumors likely to have alterations in the DNA repair mechanism (eg, CLL and other tumor types). Subjects are evaluable for efficacy if they have received at least 1 dose of study drug and have radiographic baseline. Subjects who are not evaluable for efficacy will be replaced.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumors likely to have alterations in DNA repair mechanisms, such as the BRCA and ATM pathways, or CLL, with no other standard surgical, radiation, or systemic anticancer therapies available. Subjects with CLL will be enrolled in 1 of the RP2D expansion cohorts only
* Tumor accessible for biopsies and agree to pretreatment tumor biopsy
* Measurable or evaluable disease in accordance with RECIST v 1.1 for solid tumors or Cheson´s criteria for CLL
* Male or female subjects at least 18 years of age who sign written informed consent.
* Other protocol-defined criteria could apply

Exclusion Criteria:

* Eastern Cooperative Oncology Group performance status > 1
* Prior treatment with chemotherapy, immunotherapy, hormonal therapy, with the exception of luteinizing hormone releasing hormone (LHRH) analogs, biologic therapy, any other anticancer therapy, or any other investigational agent within 28 days of the first dose of MSC2490484A (6 weeks for nitrosoureas or mitomycin C)
* Extensive prior radiotherapy on more than 30% of bone marrow reserves or prior bone marrow/stem cell transplantation within 5 years of study start. The extent of previous radiotherapy to the bone marrow will be determined by the investigator.
* Receiving medications or herbal supplements that are known to be potent inhibitors of cytochrome P450 3A4 or inducers of cytochrome P450 3A4.
* Not recovered from toxicity due to prior therapy to baseline or an AE CTCAE Grade of 1 or less (except alopecia)
* Poor vital organ function as defined in the protocol
* Significant cardiac conduction abnormalities as defined in the protocol
* Central nervous system metastases unless previously radiotherapy treated, stable by computerized tomography (CT) scan for at least 3 months without evidence of cerebral edema, and no requirements for corticosteroids or anticonvulsants
* Other protocol-defined criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-12-31 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

PRIMARY OUTCOMES:
Number of Dose limiting toxicities (DLTs) occurring in Cycle 1 | up to Day 21 of Cycle 1

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Day 1 of Cycle 1 (cycle length = 21 days)
Time to Maximum Observed Plasma Concentration (tmax) | Day 1 of Cycle 1 (cycle length = 21 days)
Minimum Observed Plasma Concentration During a Complete Dosing Interval (Cmin) | Day 1 of Cycle 1 (cycle length = 21 days)
Average Observed Plasma Concentration (Cavg) | Day 1 of Cycle 1 (cycle length = 21 days)
Fluctuation Index | Day 1 of Cycle 1 (cycle length = 21 days)
Area Under the Concentration-Time Curve From Time Zero To 24 Hours (AUC0-24) | Day 1 of Cycle 1 (cycle length = 21 days)
Area Under the Concentration-Time Curve From Time Zero To 12 Hours (AUC0-12) | Day 1 of Cycle 1 (cycle length = 21 days)
Area Under the Concentration-Time Curve From Time Zero To the Time of Last Quantifiable Concentration (AUC0-t) | Day 1 of Cycle 1 (cycle length = 21 days)
Area Under the Concentration-Time Curve From Time Zero Extrapolated To Infinity (AUC0-inf) | Day 1 of Cycle 1 (cycle length = 21 days)
Area Under the Concentration-Time Curve From Time Zero to Time tau at Steady State (AUCtau) | Day 1 of Cycle 1 (cycle length = 21 days)
Apparent Terminal Half-Life (t1/2) | Day 1 of Cycle 1 (cycle length = 21 days)
Terminal Rate Constant (λz) | Day 1 of Cycle 1 (cycle length = 21 days)
Oral Clearance (CL/f) | Day 1 of Cycle 1 (cycle length = 21 days)
Apparent Volume of Distribution During Terminal Phase (Vz/f) | Day 1 of Cycle 1 (cycle length = 21 days)
Apparent Volume of Distribution at Steady State (Vss/f) | Day 1 of Cycle 1 (cycle length = 21 days)
Accumulation Ratio for Area Under The Concentration-Time Curve (Racc[AUC]) | Day 1 of Cycle 1 (cycle length = 21 days)
Accumulation Ratio for Maximum Concentration (Racc[Cmax]) | Day 1 of Cycle 1 (cycle length = 21 days)
Best overall response rate | Time from first dose to disease progression or death, whichever occurs first, assessed until 12 weeks after last patient treated
Clinical benefit rate defined as the proportion of subjects with CR, PR, or stable disease at Week 12 | Week 12
Progression-free survival time (PFS) | Time from first dose to disease progression or death, whichever occurs first, assessed until 12 weeks after last patient treated

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (7):
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - UZ Leuven, Leuven
- Denmark (2):
  - Rigshospitalet - Onkologisk KFE, Copenhagen
  - Herlev Hospital University of Copenhagen, Herlev
- Netherlands (3):
  - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - VU Medisch Centrum - Dept of Medical Oncology, Amsterdam
  - Erasmus Medisch Centrum - Parent, Rotterdam

REFERENCES:
- [Derived] van Bussel MTJ, Awada A, de Jonge MJA, Mau-Sorensen M, Nielsen D, Schoffski P, Verheul HMW, Sarholz B, Berghoff K, El Bawab S, Kuipers M, Damstrup L, Diaz-Padilla I, Schellens JHM. A first-in-man phase 1 study of the DNA-dependent protein kinase inhibitor peposertib (formerly M3814) in patients with advanced solid tumours. Br J Cancer. 2021 Feb;124(4):728-735. doi: 10.1038/s41416-020-01151-6. Epub 2020 Nov 24. PMID 33230210